CLINICAL TRIAL: NCT06803446
Title: Effets du Rythme Circadien Sur la régulation glycémique Lors d'Exercices modérés Continus et Intermittents Intenses Chez Des Adolescents Vivant Avec le diabète de Type 1
Brief Title: Effects of Circadian Rhythm on Glycemic Regulation During Continuous Moderate Exercise and Intense Intermittent Disease in Adolescents Living With Type 1 Diabetes
Acronym: CHRONODIAB1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: D2024-05
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: adolescents; type 1 diabetes; glycemic regulation; circadian rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: 4 randomized handovers performed (on different days with meal/snack)previous standardized:
  * Continuous exercise on ergocycle in the morning
  * Continuous exercise on ergocycle in the afternoon
  * Intermittent exercise on ergocycle in the morning
  * Intermittent exercice on ergocycle in the afternoon
Masking Description: It is not possible to do a trial in blind or double blind because the moment of the day and the exercice modality can not be hidden, however the results analysis will be assessed in blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Continuous - morning (Experimental): Continuous exercise on ergocycle in the morning
- Continuous - afternoon (Experimental): Continuous exercise on ergocycle in the afternoon
  Interventions: Other: physical test
- Intermittent - morning (Experimental): Intermittent exercise on ergocycle in the morning
- Intermittent - afternoon (Experimental): Intermittent exercice on ergocycle in the afternoon
  Interventions: Other: physical test

INTERVENTIONS:
Other: physical test — continuous and intermittent exercise on cycloergometer
  Arms: Continuous - afternoon; Intermittent - afternoon

SUMMARY:
Interventional research with minimal risks and constraints on the effects of circadian rhythm on glycemic regulation during intense moderate, continuous and intermittent exercise in adolescents living with type 1 diabetes

DETAILED DESCRIPTION:
Single-center, randomized, controlled study in adolescents living with type 1 diabetes. This study aims to evaluate the effect of exercise timing (morning vs. afternoon) and exercise type (continuous vs. intermittent) on blood glucose levels during and after exercise, as well as to assess the effect of exercise timing (morning vs. afternoon) and type of exercise (continuous vs. intermittent) on blood glucose during and after exercise

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10 to 16;
* Living with type 1 diabetes for at least 1 year with HbA1c less than or equal to 12%;
* Socially insured ;
* Having given their written consent to participate in the research, as well as that of their legal guardians;
* Willing to comply with all research procedures and duration.

Exclusion Criteria:

* Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate less than 40 ml/min), neuropathy or severe proliferative retinopathy as assessed by the investigator;
* Recent acute macrovascular event (< 3 months), e.g. acute coronary syndrome or cardiac surgery;
* Abnormal blood picture and/or anemia;
* Current pregnancy;
* Other serious medical condition likely to interfere with study participation or ability to complete exercise periods in the judgment of the investigator (e.g., orthopedic limitation);
* Inability to receive informed information;
* Inability to participate in the entire study;
* Lack of social security coverage;
* Refusal to sign the consent form.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Comparison of glycemic variation between the 4 conditions | 1 year 10 months september 2026
  Observation of time in target, time in hypoglycemia and time in hyperglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasport, Loos, Nord, France

IPD SHARING:
Plan to Share IPD: No